CLINICAL TRIAL: NCT04353908
Title: The Role of Collagen in the Rehabilitation of Peripheral Paralysis of the Facial Nerve
Brief Title: Collagen Treatment in Facial Nerve Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uniter Onlus (Other)
Collaborators: University of Rome Tor Vergata (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UniterCPF
Record Dates: First submitted 2020-04-16; First posted 2020-04-21 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Facial Nerve Palsy
Keywords: Facial nerve palsy; Kabat method; Collagen injections; Electromyography
MeSH Terms: conditions — Bell Palsy | interventions — Rehabilitation; Collagen

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- kabat (Active Comparator): Rehabilitation will be started in both groups of patients and it will be carried out according to Kabat et al., i.e. a proprioceptive neuromuscular facilitation procedure, twice a week for 8 weeks, by an experienced physioptherapist
  Interventions: Procedure: Rehabilitation
- collagen injection (Experimental): Injections of an equally-balanced solution of MD Neural, MD Matrix and MD Muscle (Guna S.p.a., Milan-Italy), containing collagen of porcine origin, will be administered subcutaneously after applying lidocaine/prilocaine cream on the affected side, by a skilled otonaryngologist in the field of injection treatments, twice a week for 8 weeks
  Interventions: Procedure: Rehabilitation; Procedure: Collagen Injection

INTERVENTIONS:
Procedure: Rehabilitation — The Kabat procedure consists of facilitating the voluntary response of an impaired muscle through a global pattern of an entire muscular section which undergoes resistance. This method considers that harmony, coordination and optimal strength of body movements mainly depend upon the fact that they are performed following diagonal lines with respect to the sagittal axis of the body, thus implying a 'rotational' effect. It will performed twice a week for 8 weeks
  Other Names: Kabat procedure
Procedure: Collagen Injection — With an insulin-type syringe and 30-gauge needle, a bolus of about 0.4 cc per point of the collagen solution will be injected in the orbicularis oculi muscle 1 cm outside the orbital rim and 0.5 cm superior and inferior to the first injection point, respectively, and in the orbicularis oris muscle, where the 2 injection points are on the border between the pars peripheralis and pars marginalis, located about 5 mm above the superior and inferior vermilion, respectively
  Arms: collagen injection

SUMMARY:
To test the effectiveness of a collagen-based treatment for patients complaining of long standing facial nerve axonotmesis, who are following a proprioceptive neuromuscular facilitation protocol (Kabat method), compared to a group only undergoing the Kabat method.

DETAILED DESCRIPTION:
Objective: To test the effectiveness of a collagen-based treatment for patients complaining of long standing facial nerve axonotmesis, who are following a proprioceptive neuromuscular facilitation protocol (Kabat method), compared to a group only undergoing the Kabat method.

Methods: Patients undergoing both procedures will be compared, after randomization, to matched patients undergoing only Kabat procedure after 8 weeks of treatment. The outcomes will be electromyographic findings, validated questionnaires (Facial Disability Index, FDI) and clinical grading (House-Brackmann, HB). A correlation analysis will be performed between pre-/post-treatment diﬀerences (Δ) in outcome and clinical-demographic measures.

ELIGIBILITY:
Inclusion Criteria:

* patients with a medical diagnosis of long-term unilateral peripheral axonotmesis of the facial nerve

Exclusion Criteria:

* patients with facial palsy caused by central nerve disease;
* patients with a history of recurrent facial palsy;
* patients with a facial skin disease hampering the possibility of injecting the drug; - patients with difficulty in moving their face due to previous plastic surgery or facial surgery;
* patients with systemic diseases that can affect facial electromyography;
* patients deemed inappropriate by the researchers.
* patients with a history of hypersensitivity to any collagen solution constituent or showing pregnancy, lactation, neuromuscular junction disorders (myastenia gravis), peripheral motor neuropathies, or active infections will be also excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
duration of voluntary activity | 2 months
  An electromyography coaxial needle examination will be performed on the orbicularis oculi and orbicularis oris to evaluate the electrical alteration of these muscles. These muscles will be examined at rest and during voluntary activity in terms of msec of duration of voluntary activity

SECONDARY OUTCOMES:
Facial asymmetry | 2 months
  Static and dynamic facial asymmetry will be evaluated and manually tested on the muscle strength of the frontalis, corrugator, orbicularis oculi, zigomaticus, caninus, platysma and orbicularis oris muscles. These clinical findings will be classified and recorded according to the House-Brackmann (HB) scale, ranging from 1 (normal) to 6 (severe dysfunction).
Subjective facial disability | 2 months
  The Facial Disability Index (FDI) is a 10-item self-administered questionnaire with 2 subscale scores: 5 items concern the physical function subscale, and 5 items concern the social/well-being function subscale. Each item is rated on a 6-point scale, ranging from severe disability to absence of disability. Both subscales are transformed to a score on a 100 point scale, with 100 indicating unimpaired physical or social/wellbeing function. All questions referred to the preceding month.

CONTACTS AND LOCATIONS:
Locations (1):
- UNITER ONLUS for balance and rehabilitation research, Guidonia, Rome, Italy

REFERENCES:
- [Background] Lindsay RW, Robinson M, Hadlock TA. Comprehensive facial rehabilitation improves function in people with facial paralysis: a 5-year experience at the Massachusetts Eye and Ear Infirmary. Phys Ther. 2010 Mar;90(3):391-7. doi: 10.2522/ptj.20090176. Epub 2010 Jan 21. PMID 20093325
- [Background] Hg Beurskens C, Al Burgers-Bots I, W Kroon D, Ab Oostendorp R. Literature review of evidence based physiotherapy in patients with facial nerve paresis. J Jpn Phys Ther Assoc. 2004;7(1):35-9. doi: 10.1298/jjpta.7.35. PMID 25792936
- [Background] Barbara M, Antonini G, Vestri A, Volpini L, Monini S. Role of Kabat physical rehabilitation in Bell's palsy: a randomized trial. Acta Otolaryngol. 2010;130(1):167-72. doi: 10.3109/00016480902882469. PMID 19430987
- [Background] Cao J, Xiao Z, Jin W, Chen B, Meng D, Ding W, Han S, Hou X, Zhu T, Yuan B, Wang J, Liang W, Dai J. Induction of rat facial nerve regeneration by functional collagen scaffolds. Biomaterials. 2013 Jan;34(4):1302-10. doi: 10.1016/j.biomaterials.2012.10.031. Epub 2012 Oct 31. PMID 23122676
- [Background] Martin Martin LS, Massafra U, Bizzi E, Migliore A. A double blind randomized active-controlled clinical trial on the intra-articular use of Md-Knee versus sodium hyaluronate in patients with knee osteoarthritis ("Joint"). BMC Musculoskelet Disord. 2016 Feb 22;17:94. doi: 10.1186/s12891-016-0948-4. PMID 26905565
- [Background] Grosheva M, Wittekindt C, Guntinas-Lichius O. Prognostic value of electroneurography and electromyography in facial palsy. Laryngoscope. 2008 Mar;118(3):394-7. doi: 10.1097/MLG.0b013e31815d8e68. PMID 18090862
- [Background] Teixeira LJ, Valbuza JS, Prado GF. Physical therapy for Bell's palsy (idiopathic facial paralysis). Cochrane Database Syst Rev. 2011 Dec 7;(12):CD006283. doi: 10.1002/14651858.CD006283.pub3. PMID 22161401